CLINICAL TRIAL: NCT04492891
Title: Randomized Phase IIa Clinical Trial Of Cyclosporine For The Treatment Of COVID-19(+) Non-ICU Hospital Inpatients
Brief Title: Cyclosporine For The Treatment Of COVID-19(+)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bryan Burt, MD (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor-Investigator, Bryan Burt, MD, Associate Professor, Surgery General Thoracic, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-48163
Record Dates: First submitted 2020-07-20; First posted 2020-07-30 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-06

CONDITIONS: SARS (Disease)
Keywords: COVID-19; SARS-COV-2; Corona Virus
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Disease; COVID-19 | interventions — Cyclosporine

STUDY DESIGN:
Intervention Model Description: Phase IIa clinical trial in which 75 non-ICU hospital inpatients will be randomized 2:1 to 7 days of Neoral (2.5mg/kg PO BID) + standard of care (SOC) or no CSA + SOC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A Cyclosporine (Experimental): Neoral, N=50 Patients 2.5 mg/kg PO BID 7 days
  Interventions: Drug: Cyclosporine
- Arm B Standard of Care (Other): Standard of Care Treatment, N= 25 Patients 7 days
  Interventions: Other: Standard of Care Treatment

INTERVENTIONS:
Drug: Cyclosporine — 2.5 mg/kg PO BID 7 days
  Other Names: Neoral
  Arms: Arm A Cyclosporine
Other: Standard of Care Treatment — Standard of Care Treatment, N= 25 Patients, 7 days
  Arms: Arm B Standard of Care

SUMMARY:
Phase IIa clinical trial in which 75 non-ICU hospital inpatients will be randomized 2:1 to 7 days of an oral formulation of cyclosporine, Neoral (2.5mg/kg PO BID) + standard of care (SOC) or no Neoral + SOC. The primary endpoint is disease severity based on the World Health Organization (WHO) COVID Ordinal Outcomes Scale, on day 14. Secondary endpoints include safety and changes in serum inflammatory markers.

DETAILED DESCRIPTION:
1. OBJECTIVES

   1.1 Primary Objectives

   1.1.1 To assess the effect of a 7-day course of oral cyclosporine Neoral on clinical outcome using the World Health Organization (WHO) COVID Ordinal Clinical Outcomes Scale, on day 14.

   1.2 Secondary Objectives

   1.2.1 To establish the safety of Neoral in this patient population (adverse events).

   1.2.2 To determine the effect of Neoral on serum inflammatory markers (CRP, d-dimer, ferritin, ANC (Absolute Neutrophil Count), absolute lymphocyte count, WBC, PLT (daily while inpatient and including day 14 and 28 for those discharged).

   1.2.3 To determine the effect Neoral on viral SARS-CoV2 PCR positivity from baseline (day 0 to -2) before receiving Neoral to day 14, and from baseline to day 28.

   1.2.4 To determine the effect of Neoral on survival (days 14 and 28).

   1.2.5 To determine the effect of Neoral on disease improvement (alive and free of invasive or non-invasive mechanical ventilation; days 14 and 28).

   1.2.6 To determine the effect of Neoral on proportion of those requiring invasive mechanical ventilation.

   1.2.7 To determine the effect of Neoral on incidence of deep vein thrombosis.

   1.2.8 To determine the effect of Neoral on proportion of patients discharged on day 28.

   1.2.9 To determine the effect of Neoral on time to hospital discharge.

   1.2.10 To determine the effect of Neoral on disease resolution (alive and discharged home without oxygen; days 14 and 28).
2. BACKGROUND

2.1 Study Disease(s)

Severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) is a novel coronavirus that causes coronavirus disease 2019 (COVID-19). Since initial detection of the virus, more than 10 million cases of COVID-19 have been confirmed worldwide, and COVID-19 is responsible for more than 505,500 deaths. The United States has seen over 2.5 million cases of COVID-19 and 126,000 deaths from this disease (as of June, 30, 2020). SARS-CoV-2 is efficiently transmitted from person-to-person and the World Health Organization (WHO) has declared coronavirus disease 2019 (COVID-19) to be a pandemic.

COVID-19 primarily spreads through the respiratory tract, by droplets, respiratory secretions, and direct contact. Current data suggest an incubation period of 1-14 days, in most cases 3-7 days. The virus is highly transmissible in humans and causes severe problems especially in the elderly and people with underlying chronic diseases. COVID-19 patients typically present with specific, similar symptoms, such as fever, malaise, and cough. Most adults or children infected with SARS-CoV-2 have presented with mild flu-like symptoms, but a few patients are in critical condition and rapidly develop acute respiratory distress syndrome (ARDS), respiratory failure, multiple organ failure, and death. The case fatality rate increases with the severity of illness and can reach up to 49% in critically ill patients.

Unfortunately, specific and effective therapies for COVID-19 are highly limited. Recent evidence suggest that administration of the anti-viral agent, Remdesivir, to hospital inpatients with COVID-19 decreases time to recovery from 15 to 11 days and decreases mortality at 14 days from 11.9% to 7.1%. A preliminary, unpublished analysis from a large, multicenter, randomized, open-label trial for hospitalized patients in the United Kingdom showed that patients who were randomized to receive dexamethasone had a reduced rate of mortality compared to those who received standard of care. This benefit was observed in patients with severe COVID-19 and was greatest in those who required mechanical ventilation at enrollment (RECOVERY Trial). These 2 agents are considered in the standard of care (SOC) for treating patients with COVID-19. However, additional therapies with larger effect sizes and that are administered at earlier stages to prevent progression to severe COVID-19 are critically needed.

2.1.1 IND (Investigational New Drug) Agent(s)

The PI has filed an IND with cross-reference letter from Novartis and has received a Safe to Proceed determination (IND #152065).The rationale for the proposed starting dose is based on the standard renal transplantation dose, which has a time-honored profile of safety in this population.

2.2 Rationale

Severe COVID-19. Initial reports from cases identified between February 12 to March 16 in the United States (U.S.) show rates of hospitalization for COVID-19 to be 21-31%, intensive care unit (ICU) admissions to be 5- 12%, and fatality to be 2%-3%. High-risk groups for severe COVID-19 have been identified as the elderly population and those with underlying comorbidities such as cardiovascular disease, liver disease, pulmonary disease, renal disease, and diabetes mellitus.

Severe COVID-19 results from a dysregulated hyperimmune state. Severe symptoms of COVID-19 are associated with a hyperimmune response referred to as a cytokine storm. In one study, all 41 patients with COVID-19 admitted to the hospital demonstrated elevated plasma levels of cytokines and chemokines compared with healthy volunteers that included IL (Interleukin) -1, -1R, -7, -8, -9, -10, and basic FGF2, GCSF, GMCSF, IFN-γ, IP10, MCP1, M1P1A, MIP1B, PDGF, TNF-α, and VEGF. Patients admitted to the ICU had higher levels of IL-2, IL-7, IL-10, GCSF, IP10, MCP1, MIP1A, and TNF-α than patients who did not require ICU admission. Emerging data has shown that early rapid SARS-CoV-2 replication causes massive epithelial and endothelial cell death that initiates a cytokine storm and vascular leakage, causes pyroptosis in macrophages and lymphocytes, and results in exhaustion of T cells and NK (Natural Killer) cells.

COVID-19 similarities to hemophagocytic lymphohistiocytosis (HLH). HLH is an under-recognized, hyperinflammatory syndrome characterized by a fulminant and fatal cytokine storm and multi-organ failure. In adults, HLH is most commonly triggered by viral infections and occurs in 3.7% to 4.3% cases of sepsis. Cardinal features include unremitting fever, cytopenias, and hyperferritinemia. Pulmonary involvement (including ARDS) occurs in ~50% of patients. Each of these clinical features and a highly overlapping cytokine profile is seen in severe COVID-19. This demonstrates that the clinical presentation and pathologic mechanisms of severe COVID-19 is similar to, or is HLH.

Cyclosporine (CSA) suppresses hyperimmune states. Calcineurin inhibitors such as CSA suppress the phosphatase activity of calcineurin, which results in decreased IL-2 production and IL-2 receptor expression. This interrupts a central pathway of T-cell activation and dampens T cell responses and their associated cytokine storms. CSA is approved by the FDA for three indications including 1) prophylaxis of organ rejection in kidney, liver, and heart transplants, 2) treatment of severe active rheumatoid arthritis, and 3) treatment of adult severe recalcitrant plaque psoriasis. It is critical to consider whether dampening of T-cell responses using CSA would curtail the vigor of T-cell hyperactivity in COVID-19 disease and provide an opportunity for these patients to recover.

CSA for COVID-19. Proposed is the use of the calcineurin inhibitor, CSA, for the treatment of patients with COVID-19. This is based on: 1) observations that COVID-19 disease is associated with a hyperimmune response very similar to HLH, for which treatment with CSA is effective and recommended, 2) COVID-19 is associated with dysregulated macrophage activation similar to macrophage activation syndrome (MAS) which is also therapeutically suppressed by CSA, and 3) in vitro studies demonstrating that CSA specifically inhibits the replication of coronaviruses including SARS-CoV-2 with a high degree of specificity.

CSA specifically inhibits coronavirus replication. Coronaviruses are RNA viruses with large genomes that enter host cells through binding of its transmembrane spike protein with angiotensin-converting enzyme 2 (ACE2) receptors expressed by host target cells, which is the same mechanism utilized by SARS-CoV (i.e., SARS). Cyclophilins appear to play a critical role in the replication of many viruses including coronaviruses, HIV, and hepatitis C virus. Although the exact mechanisms are not yet well understood, in vitro studies suggest that the coronavirus' nonstructural protein (Nsp) and nucleocapsid protein bind to cyclophilins, and knockdown of cyclophilin expression results in near complete inhibition of coronavirus replication. These data show that viral protein binding to cyclophilins is an important step for successful coronavirus replication, and inhibition of this interaction by CSA prevents viral replication. An important study demonstrated that CSA dominantly inhibited replication of human coronavirus 229E (HCoV-229E), mouse hepatitis virus (MHV), and SARS, and that treatment with increasing doses of CSA caused a dose-dependent decrease in SARS-CoV replication in human cells in vitro without affecting cell viability. The same group demonstrated that CSA inhibited replication of MERS-CoV without affecting cell viability of mock-infected cells. An independent group demonstrated that increasing concentrations of CSA treatment of SARS-CoV-infected human cells resulted in a dose-dependent decrease in viral replication, and inhibited the replication of other coronaviruses, including human CoV-NL63, CoV-229E, feline CoV serotypes I and II, porcine transmissible gastroenteritis virus (TGEV), avian infection bronchitis virus (IBV), and two isolates of SARS-CoV. Taken together it is proposed a dual mechanism in which (1) calcineurin inhibition by CSA inhibits the phosphorylation of NFAT-P, thus preventing the production of IL-2 and other proinflammatory cytokines, and (2) CSA inhibits viral replication of coronaviruses, likely through blockade of calcineurin, causing the inhibition of cyclophilins required for viral replication. Most recently, it was demonstrated that CSA is highly specific and effective at inhibiting SARS-CoV-2 replication in various human cells, via inhibition of Cyclophilin.

Safety of CSA in COVID-19. Since April 2020 mounting evidence from various patient populations has strongly suggested that CSA can be used safely in patients with COVID-19. It was recently demonstrated that patients with "Immune Mediated Inflammatory Diseases" (IMID) on various immunosuppressive drugs related to CSA have a "significantly reduced incidence of SARS-CoV-2 infection". It was reported no significant increase in the incidence or severity of COVID-19 disease in patients undergoing CSA therapy for Psoriasis, but rather suggested a potentially milder disease in these patients. Another study of over 4000 patients in Madrid, Spain demonstrated "a universal relationship between the use of Cyclosporine A and better outcomes" in patients with COVID-19 disease. In line with the findings from Spain, Cavagna in Italy observed that transplant patients with ongoing Calcineurin Inhibitor therapy developed only mild symptoms of COVID-19 disease and concluded that "Calcineurin inhibitor-based immunosuppressive regimens appear safe" in COVID-19 disease and should not be discontinued. These recent clinical outcomes data suggest that the use of CSA in patients with COVID-19 is safe and potentially effective.

2.3 Correlative Studies Background

Correlative studies in this protocol are included as secondary endpoints and are based on: 1) serum inflammatory markers used clinically as biomarkers to monitor the severity of COVID-19 (CRP, d-dimer, ferritin, ANC, absolute lymphocyte count, WBC (White Blood Cells), PLT), and 2) SARS-CoV-2 viral load by a clinical PCR (Polymerase Chain Reaction) test.

6. TREATMENT AND/OR IMAGING PLAN

6.1 Agent Administration

Treatment will be administered on an inpatient basis.

Arm A Regimen Description Agent Neoral, Investigational, Generic Acceptable, N=50 Patients 2.5 mg/kg PO BID 7 days

Arm B Regimen Description Agent None*, N= 25 Patients 7 days

*Note: The PI has undertaken thorough discussions with the sponsor and generation of placebo capsules is not feasible for the timing of this study.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 Laboratory-confirmed SARS-CoV-2 infection within the past 10 days.

3.1.2 Patients admitted to non-ICU hospital floors or in an emergency department awaiting admission to a non-ICU hospital bed.

3.1.3 WHO COVID Scale Score 4 (Oxygen by mask or nasal prongs or WHO COVID Scale Score 5 (non-invasive ventilation or high-flow oxygen).

3.1.4 Age 18 to 90 years old.

3.1.5 ECOG (Eastern Cooperative Oncology Group) performance status ≤2 (see Appendix A).

3.1.6 Patients receiving or who have received standard of care therapy for COVID-19 can be included. This includes Remdesivir, Dexamethasone (or other steroids), and convalescent plasma.

3.1.7 Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

3.2.1 Allergy and/or hypersensitivity to CSA.

3.2.2 GFR<30 mL/min.

3.2.3 ALT (Alanine transaminase) or AST (Aspartate transaminase) >3X upper limits of normal.

3.2.4 Resistant hypertension (BP>140/90 mm Hg despite adherence to maximal doses of three antihypertensive agents).

3.2.5 Active bacterial or mycobacterial infection.

3.2.6 Pregnant and/or nursing patients. 3.2.7 Participation in a COVID-19 therapeutic drug trial.

3.2.8 Patients who have received or who are receiving anti-viral medications including hydroxychloroquine will not be excluded.

3.2.9 Patients with psychiatric illness/social situations that would limit compliance with study requirements.

3.2.10 Total cholesterol is < 100 (increased risk of seizure)

3.2.11 Concomitant dosing with Tacrolimus is a relative contraindication (increases overall immunosuppression and decrease seizure threshold

3.2.12 Concomitant malignancy is a relative contraindication (Neoral can increase susceptibility to development of neoplasia)

3.2.13 Inability to swallow oral medication

3.2.14 Treatment with immunomodulators or immunosuppressant drugs, including but not limited to IL-6 inhibitors, TNF inhibitors, anti-IL-1 agents, and JAK inhibitors.

3.2.15 Investigational Antiviral agents

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Burt, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one institution between November 2020 and October 2021. The first participant enrolled on November 23, 2020, and the last participant enrolled on October 12, 2021.
Pre-assignment Details: Due to the decline of COVID-19 cases which led to slow accrual, the study was closed to enrollment on April 6, 2022. For this reason, the total number of participants reported in the Brief Summary and the enrollment number of participants have a discrepancy.
Groups:
- Arm A Cyclosporine: Participants received Neoral 2.5mg/kg PO BID, based on the renal transplant dose for 7 days.
  Neoral is an oral formulation of cyclosporine.
- Arm B Standard of Care: Participants received standard of Care Treatment(no taking Neoral) for 7 days
Period: Overall Study
Arm/Group | Arm A Cyclosporine | Arm B Standard of Care
Started (Due to the decline of COVID-19 cases which led to slow accrual, the study was closed to enrollment on April 6, 2022. For this reason, the total number of participants reported in the Arm/Group Description and the number of participants who started in the Participant Flow of the Result Section have a discrepancy.) | 30 | 17
Completed (Due to the decline of COVID-19 cases which led to slow accrual, the study was closed to enrollment on April 6, 2022. For this reason, the total number of participants reported in the Arm/Group Description and the number of participants who completed in the Participant Flow of the Result Section have a discrepancy.) | 30 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A Cyclosporine | Arm B Standard of Care | Total
Number analyzed (Participants) | 30 | 17 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (14.8) | 59.8 (14.9) | 59.8 (14.7)
Age, Customized [Count of Participants; unit: Participants]
  Age category: < 60 years | 14 | 8 | 22
  Age category: >= 60 years | 16 | 9 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 18 | 10 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 14
  Not Hispanic or Latino | 20 | 12 | 32
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 20 | 12 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
WHO score - score 4 [Count of Participants; unit: Participants] — WHO COVID-19 clinical severity scale range is from 0 (uninfected) to 8 (death). WHO score 4 is in Hospitalized Mild disease status which a patient needs Oxygen by mask or nasal prongs.
  Participants | 30 | 17 | 47
Comorbidity [Count of Participants; unit: Participants] — if participants had at least one of the following- hypertension, coronary artery disease, congestive heart failure, or diabetes, then comorbidity is "Presence" otherwise "absence"
  Participants
    Absence | 9 | 6 | 15
    Presence | 21 | 11 | 32

OUTCOME MEASURES:

1. Primary Outcome: WHO(World Health Organization) COVID-19 Clinical Severity Scale
Description: WHO(World Health Organization) COVID-19 clinical severity scale. Score 0-9. 0=Uninfected, 8=Death.
Time Frame: on day 14
Population: WHO scores were obtained during ± 3 days on each planned day 14. If no WHO score is available on the planned day because of early discharge, the last WHO score was used for analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Arm A Cyclosporine | Arm B Standard of Care
Number analyzed (Participants) | 30 | 17
units on a scale | 2 [0 to 3] | 2 [1 to 2]

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Arm A Cyclosporine | Arm B Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/17
Other Adverse Events (participants affected / at risk) | 13/30 | 1/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Cyclosporine (N=30) | Arm B Standard of Care (N=17)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) — Chest pain - cardiac
Death NOS (General disorders) | 1 (1) | 0 (0) — Death NOS
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) — Alanine aminotransferase increased
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) — Aspartate aminotransferase increased
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Cyclosporine (N=30) | Arm B Standard of Care (N=17)
Chest pain - cardiac (Cardiac disorders) | 4 (4) | 0 (0) — Chest pain - cardiac
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Ear pain
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Constipation
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Nausea
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Vomiting
Sepsis (Infections and infestations) | 1 (1) | 0 (0) — Sepsis
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) — Alanine aminotransferase increased
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) — Aspartate aminotransferase increased
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0) — Investigations - Other, specify
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Back pain
Headache (Nervous system disorders) | 1 (1) | 0 (0) — Headache
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) — Confusion
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) — Acute kidney injury
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Adult respiratory distress syndrome
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Hypoxia
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Respiratory, thoracic and mediastinal disorders - Other, specify
Hypertension (Vascular disorders) | 0 (0) | 1 (1) — Hypertension

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT04492891/Prot_SAP_000.pdf